CLINICAL TRIAL: NCT06601907
Title: Researching the Effectiveness of a Alivis, a Digital Health Application for Borderline Personality Disorder: a Randomized Controlled Trial
Brief Title: Researching the Effectiveness of a Alivis, a Digital Health Application for Borderline Personality Disorder
Acronym: REVALDI-BPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: Zentrum fÃ¼r Integrative Psychiatrie (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: alivis RCT 2024
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Borderline Personality Disorder (BPD)
Keywords: Digital Intervention; Borderline Personality Disorder; RCT; Dialectical Behavior Therapy
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alivis + TAU (Experimental): Participants in the intervention group will receive access to alivis in addition to treatment as usual (TAU) for 12 months.
  Interventions: Behavioral: alivis
- TAU (No Intervention): Participants in the control group will receive access to treatment as usual (TAU) only. They will receive access to alivis after their last study visit (T3; 12 months after randomization).

INTERVENTIONS:
Behavioral: alivis — alivis is an interactive online program for independent use by users with Borderline Personality Disorder. It focuses on recognized treatment elements from Dialectical Behavior Therapy, Schema Therapy, Acceptance and Commitment Therapy, and Mindfulness Self-Compassion Therapy.
  Arms: alivis + TAU

SUMMARY:
This randomized controlled trial (RCT) with 470 patients diagnosed with Borderline Personality Disorder (BPD) aims to investigate the effectiveness of the unguided digital therapeutic alivis for patients with BPD as defined in DSM-5. Inclusion criteria are: male, female or non-binary, age 18-65 years, diagnosis of BPD (confirmed by SCID-5-PD), borderline severity score (cut-off) of ≥ 1.07 on the Borderline Symptoms List 23 (BSL-23), stable treatment (psychotherapy, medication, no treatment, …) for at least 30 days at the time of inclusion, consent to emergency plan for suicidal crises, consent to participation, and sufficient German language skills. Exclusion criteria are: Plans to change in treatment (psychotherapy, medication, …) in the upcoming 6 months after inclusion, comorbid diagnosis of substance use disorder or lifetime diagnosis of psychotic disorder, physical condition that can cause severe psychiatric symptoms, acute decompensation of mental health, BMI <15, and prior use of the digital intervention priovi.

Patients will be randomized and allocated to either an intervention group, in which they will receive access to alivis in addition to treatment as usual (TAU; n=235), or to a control group, in which they will receive access to TAU (n=235).

The primary endpoint will be BPD symptoms with three months post-allocation (T1) being the primary timepoint for assessment of effectiveness. Six (T2) and twelve (T3) months post-allocation will be used as follow-up assessment of endpoints. Secondary endpoints will be depressive symptoms, anxiety symptoms, costs caused due to the patient's BPD, social functioning, health-related quality of life, and patient activation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BPD
* Borderline severity score (cut-off) of ≥ 1.07 on the BSL-23
* Stable treatment (e.g., psychotherapy, medication, no treatment) for at least 30 days at the time of inclusion
* Consent to emergency plan for suicidal crises
* Consent to participation
* Sufficient knowledge of the German language

Exclusion Criteria:

* Plans to change treatment (e.g., psychotherapy, medication) in the upcoming 6 months after inclusion
* Comorbid diagnosis of substance use disorder
* Lifetime diagnosis of psychotic disorder like schizophrenia or schizoaffective disorder (except non-transitory paranoid ideas that can be concomitant with BPD and in which the ability to test reality is mostly preserved)
* Diagnosis of a physical condition that can cause serious psychiatric symptoms
* Acute decompensation of mental health symptoms, e.g. acute manic state or acute suicidality
* BMI < 15
* Current psychiatric day-care or inpatient treatment
* Prior use of the digital intervention priovi

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Borderline Symptoms List 23 (BSL-23) | T1 (3 months after randomization)
  The BSL-23 is a 23-item PROM with good psychometric properties that was validated and tested for reliability in a representative German sample (test-retest reliability r = .82, p < 0.0001; α = 0.94-0.97; high correlation of total score with general psychological burden and depression) to assess the typical symptomatology and severity of BPD. It refers to the last week and has a range from 0 = "not at all" to 4 = "very strong". Its single factor structure was optimized to reflect levels and changes in severity of BPD-symptomatology based on a mean score.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | T1 (3 months after randomization)
  The PHQ-9 is the 9-item depression module from the full PHQ with comparable sensitivity and specificity, and includes the 9 criteria upon which the diagnosis of DSM-IV depressive disorders is based. Rating is done on a 4-point Likert scale ranging 0 = "not at all" to 3 = "nearly every day". As a severity measure, scores range from 0 to 27 and represent: mild (&lt;5), moderate (5-9), moderately severe (10-14), and severe depression (≥15). According to several studies, the German version can be considered reliable regarding psychometric standards.
Generalized Anxiety Disorder Assessment 7 (GAD-7) | T1 (3 months after randomization)
  This self-administered patient questionnaire is used as a screening tool and severity measure for generalized anxiety disorder (GAD). Studies report good reliability, as well as criterion, construct, factorial, and procedural validity. The GAD-7 is scored on a Likert scale ranging from 0 = "not at all" via 1 = "several days" and 2 = "more than half the days" to 3 = "nearly every day", yielding a sum score ranging from 0-21. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Costs caused due to the patients BPD | T1 (3 months after randomization)
  Costs caused due to BPD will be assessed with a self-compiled instrument assessing inpatient and outpatient treatment, support from friends, family and professional services, contacts with members of the judicial authorities and public security, medication, sick leave, and physician/therapist visits during work time.
Work and Social Adjustment Scale (WSAS) | T1 (3 months after randomization)
  The WSAS is a 5-item self-report scale to measure social functioning in regard to physical, mental and social health as well as age group referenced competence for performance. The PROM has good psychometric properties with good criterion validity, good sensitivity and strong internal consistency (α = 0.89). Individual items address work, home management, social leisure, private leisure and relationships. Each item is rated on a 9-point Likert scale from 0 = "not at all impaired" to 8 = "very severely impaired". The total score has a range of 0-40, with lower scores denoting less disability.
Patient Activation Measure (PAM-13) | T1 (3 months after randomization)
  The PAM-13 assesses patients' active participation in their medical care using 13 items. Items are answered using a Likert scale ranging from 1 = "strongly disagree" to 4 = "agree strongly", yielding a total score between 13 and 52. The German version of the PAM-13, the PAM-13-G, is validated and demonstrates good psychometric properties, including a good internal consistency of Cronbach's α = 0.84.
Assessment of Quality of Life 8 Dimensions (AQoL-8D) | T1 (3 months after randomization)
  The AQoL-8D is a health-related quality-of-life questionnaire consisting of 35 items forming eight health dimensions: independent living, happiness, mental health, coping, relationships, self worth, pain, senses. Validation of the AQoL-8D assessing health-related quality of life showed good psychometric properties in a German patient sample, including excellent reliability (Cronbach's α = 0.96) and construct validity (strong correlation with the SF-36, r = .81). The AQoL-8D score ranges from 0-100; higher scores indicating higher quality of life.

OTHER OUTCOMES:
Assessment of Quality of Life 8 Dimensions (AQoL-8D) | T2 (6 months after randomization); T3 (12 months after randomization)
  The AQoL-8D is a health-related quality-of-life questionnaire consisting of 35 items forming eight health dimensions: independent living, happiness, mental health, coping, relationships, self worth, pain, senses. Validation of the AQoL-8D assessing health-related quality of life showed good psychometric properties in a German patient sample, including excellent reliability (Cronbach's α = 0.96) and construct validity (strong correlation with the SF-36, r = .81). The AQoL-8D score ranges from 0-100; higher scores indicating higher quality of life.
Patient Activation Measure (PAM-13) | T2 (6 months after randomization); T3 (12 months after randomization)
  The PAM-13 assesses patients' active participation in their medical care using 13 items. Items are answered using a Likert scale ranging from 1 = "strongly disagree" to 4 = "agree strongly", yielding a total score between 13 and 52. The German version of the PAM-13, the PAM-13-G, is validated and demonstrates good psychometric properties, including a good internal consistency of Cronbach's α = 0.84.
Work and Social Adjustment Scale (WSAS) | T2 (6 months after randomization); T3 (12 months after randomization)
  The WSAS is a 5-item self-report scale to measure social functioning in regard to physical, mental and social health as well as age group referenced competence for performance. The PROM has good psychometric properties with good criterion validity, good sensitivity and strong internal consistency (α = 0.89). Individual items address work, home management, social leisure, private leisure and relationships. Each item is rated on a 9-point Likert scale from 0 = "not at all impaired" to 8 = "very severely impaired". The total score has a range of 0-40, with lower scores denoting less disability.
Costs caused due to the patients BPD | T2 (6 months after randomization); T3 (12 months after randomization)
  Costs caused due to BPD will be assessed with a self-compiled instrument assessing inpatient and outpatient treatment, support from friends, family and professional services, contacts with members of the judicial authorities and public security, medication, sick leave, and physician/therapist visits during work time.
Generalized Anxiety Disorder Assessment 7 (GAD-7) | T2 (6 months after randomization); T3 (12 months after randomization)
  This self-administered patient questionnaire is used as a screening tool and severity measure for generalized anxiety disorder (GAD). Studies report good reliability, as well as criterion, construct, factorial, and procedural validity. The GAD-7 is scored on a Likert scale ranging from 0 = "not at all" via 1 = "several days" and 2 = "more than half the days" to 3 = "nearly every day", yielding a sum score ranging from 0-21. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Patient Health Questionnaire 9 (PHQ-9) | T2 (6 months after randomization); T3 (12 months after randomization)
  The PHQ-9 is the 9-item depression module from the full PHQ with comparable sensitivity and specificity, and includes the 9 criteria upon which the diagnosis of DSM-IV depressive disorders is based. Rating is done on a 4-point Likert scale ranging 0 = "not at all" to 3 = "nearly every day". As a severity measure, scores range from 0 to 27 and represent: mild (&lt;5), moderate (5-9), moderately severe (10-14), and severe depression (≥15). According to several studies, the German version can be considered reliable regarding psychometric standards.
Borderline Symptoms List 23 (BSL-23) | T2 (6 months after randomization); T3 (12 months after randomization)
  The BSL-23 is a 23-item PROM with good psychometric properties that was validated and tested for reliability in a representative German sample (test-retest reliability r = .82, p &lt; 0.0001; α = 0.94-0.97; high correlation of total score with general psychological burden and depression) to assess the typical symptomatology and severity of BPD. It refers to the last week and has a range from 0 = "not at all" to 4 = "very strong". Its single factor structure was optimized to reflect levels and changes in severity of BPD-symptomatology based on a mean score.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Philipp Klein, Prof. Dr., Principal Investigator — Universität zu Lübeck, Zentrum für Integrative Psychiatrie
Locations (1):
- GAIA, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No